CLINICAL TRIAL: NCT03134807
Title: The Very Old Intensive Care Patient: A Multinational Prospective Observation Study
Acronym: VIP1
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Hans Flaatten, Professor and senior ICU consultant, University of Bergen
Other Study IDs: ESICM VIP1
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Critical Illness; Old Age; Debility; Survival
MeSH Terms: conditions — Critical Illness; Frailty | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Admission of elderly ICU patients (≥80): All consecutibve admission in 3 month period or 20 pateints
  Interventions: Other: Observation prospective

INTERVENTIONS:
Other: Observation prospective — No intervention
  Other Names: Observation and registration of data

SUMMARY:
* The primary aim is to document the incidence and short-term outcome of the elderly ICU patient (≥ 80 years) using a multicentre, multi national approach
* The secondary aim is to investigate the properties of a simple frailty index in this cohort, and in particular if this is an instrument that can be used in resource and outcome prediction in this group
* To create hypothesis for further studies, in particular on various outcome prediction

DETAILED DESCRIPTION:
The investigators have chosen to use a prospective registration of routinely collected data in this ICU population. The study is mainly European based, but will also allow for ICUs outside Europe to participate.

20 consecutive ICU admission in patients ≥ 80 years of age will be collected OR all patients ≥ 80 years in a three months' period (whatever comes first).

Data are collected electronically through an e-CRF and with baseline documentation of the ICU. The database is located in Denmark, at the Department of Epidemiology, University of Aarhus (http://vip1study.com/) . Each ICU will only have access through the database of their own patients, and patient ID is not registered (Names, birth-date or social security numbers) so it is in that sense anonymous.

Even with de-identified data, most countries must seek necessary consent from the authorities to collect such data, and hence there will be a period between ICU recruitment (starting April 2016) and patient recruitment (October 1. 2016) to allow for this to be done prior to study start.

The goal is to recruit at least 100 ICUs which will give data from approximately 2000 elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* All admissions in the group

Exclusion Criteria:

* None

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Critical ill elderly patients admitted to an ICU
Sampling Method: Non-Probability Sample
Enrollment: 5132 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Survival | 30 days
  ICU and 30 days
Frailty | Pre admission
  Clinical Frailty Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hans Flaatten, Prof, Principal Investigator — University of bergen; ESICM
Locations (1):
- General ICU, KSK; Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beil M, van Heerden PV, de Lange DW, Szczeklik W, Leaver S, Guidet B, Flaatten H, Jung C, Sviri S, Joskowicz L. Contribution of information about acute and geriatric characteristics to decisions about life-sustaining treatment for old patients in intensive care. BMC Med Inform Decis Mak. 2023 Jan 6;23(1):1. doi: 10.1186/s12911-022-02094-z. PMID 36609257
- [Derived] Bruno RR, Wernly B, Kelm M, Boumendil A, Morandi A, Andersen FH, Artigas A, Finazzi S, Cecconi M, Christensen S, Faraldi L, Lichtenauer M, Muessig JM, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Leaver S, Boulanger C, Walther S, Schefold JC, Joannidis M, Nalapko Y, Elhadi M, Fjolner J, Zafeiridis T, De Lange DW, Guidet B, Flaatten H, Jung C; VIP2 study group. Management and outcomes in critically ill nonagenarian versus octogenarian patients. BMC Geriatr. 2021 Oct 19;21(1):576. doi: 10.1186/s12877-021-02476-4. PMID 34666709
- [Derived] Fronczek J, Polok K, de Lange DW, Jung C, Beil M, Rhodes A, Fjolner J, Gorka J, Andersen FH, Artigas A, Cecconi M, Christensen S, Joannidis M, Leaver S, Marsh B, Morandi A, Moreno R, Oeyen S, Agvald-Ohman C, Bollen Pinto B, Schefold JC, Valentin A, Walther S, Watson X, Zafeiridis T, Sviri S, van Heerden PV, Flaatten H, Guidet B, Szczeklik W; VIP1; VIP2 study group. Relationship between the Clinical Frailty Scale and short-term mortality in patients >/= 80 years old acutely admitted to the ICU: a prospective cohort study. Crit Care. 2021 Jul 1;25(1):231. doi: 10.1186/s13054-021-03632-3. PMID 34210358
- [Derived] Wernly B, Beil M, Bruno RR, Binnebossel S, Kelm M, Sigal S, van Heerden PV, Boumendil A, Artigas A, Cecconi M, Marsh B, Moreno R, Oeyen S, Bollen Pinto B, Szczeklik W, Leaver S, Walther SM, Schefold JC, Joannidis M, Fjolner J, Zafeiridis T, de Lange D, Guidet B, Flaatten H, Jung C; VIP2 study group. Provision of critical care for the elderly in Europe: a retrospective comparison of national healthcare frameworks in intensive care units. BMJ Open. 2021 Jun 3;11(6):e046909. doi: 10.1136/bmjopen-2020-046909. PMID 34083342
- [Derived] Wernly B, Bruno RR, Kelm M, Boumendil A, Morandi A, Andersen FH, Artigas A, Finazzi S, Cecconi M, Christensen S, Faraldi L, Lichtenauer M, Muessig JM, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Niederseer D, Valentin A, Watson X, Leaver S, Boulanger C, Walther S, Schefold JC, Joannidis M, Nalapko Y, Elhadi M, Fjolner J, Zafeiridis T, De Lange DW, Guidet B, Flaatten H, Jung C. Sex-specific outcome disparities in very old patients admitted to intensive care medicine: a propensity matched analysis. Sci Rep. 2020 Oct 29;10(1):18671. doi: 10.1038/s41598-020-74910-3. PMID 33122713
- [Derived] Jung C, Wernly B, Muessig JM, Kelm M, Boumendil A, Morandi A, Andersen FH, Artigas A, Bertolini G, Cecconi M, Christensen S, Faraldi L, Fjolner J, Lichtenauer M, Bruno RR, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Zafeiridis T, De Lange DW, Guidet B, Flaatten H; VIP1 study group. Electronic address: hans.flaatten@uib.no. A comparison of very old patients admitted to intensive care unit after acute versus elective surgery or intervention. J Crit Care. 2019 Aug;52:141-148. doi: 10.1016/j.jcrc.2019.04.020. Epub 2019 May 2. PMID 31055187
- [Derived] Muessig JM, Nia AM, Masyuk M, Lauten A, Sacher AL, Brenner T, Franz M, Bloos F, Ebelt H, Schaller SJ, Fuest K, Rabe C, Dieck T, Steiner S, Graf T, Janosi RA, Meybohm P, Simon P, Utzolino S, Rahmel T, Barth E, Schuster M, Kelm M, Jung C. Clinical Frailty Scale (CFS) reliably stratifies octogenarians in German ICUs: a multicentre prospective cohort study. BMC Geriatr. 2018 Jul 13;18(1):162. doi: 10.1186/s12877-018-0847-7. PMID 30005622
- [Derived] Flaatten H, De Lange DW, Morandi A, Andersen FH, Artigas A, Bertolini G, Boumendil A, Cecconi M, Christensen S, Faraldi L, Fjolner J, Jung C, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Zaferidis T, Guidet B; VIP1 study group. The impact of frailty on ICU and 30-day mortality and the level of care in very elderly patients (>/= 80 years). Intensive Care Med. 2017 Dec;43(12):1820-1828. doi: 10.1007/s00134-017-4940-8. Epub 2017 Sep 21. PMID 28936626